CLINICAL TRIAL: NCT00131040
Title: Investigation of Leukocyte Trafficking Into Skin Blisters During Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FS/03/065/15951
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2005-08

CONDITIONS: Ischemic Heart Disease; Angina Pectoris
Keywords: Cardiopulmonary; Surgery; leukocyte; inflammation; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris; Inflammation | interventions — Aprotinin

INTERVENTIONS:
Drug: Aprotinin

SUMMARY:
The purpose of this study was to see if the heart-lung machine involved in cardiac surgery increases the movement of activated white blood cells from the bloodstream into the patient's tissues and also to see if aprotinin usage during surgery reduces this effect.

DETAILED DESCRIPTION:
It has long been known that exposure of blood to the heart-lung bypass machine can trigger a whole-body inflammatory response in cardiac surgery patients that is linked to activation of circulating white blood cells. The investigators propose to use a technique to track the movement of white blood cells into the skin of patients during bypass surgery. The skin blisters will be elicited by application of the blistering agent cantharidin to the forearm of volunteer patients. This will allow the investigators to study the activation state of white blood cells that enter tissues during bypass surgery and to determine whether aprotinin has any beneficial effect with regards to inflammatory status of these cells.

The investigators propose that white blood cell trafficking into the blisters will increase following the use of the heart-lung machine and that the effect of aprotinin will be to ablate this.

ELIGIBILITY:
Inclusion Criteria:

* Primary elective coronary artery bypass surgery

Exclusion Criteria:

* Emergent, urgent or re-do surgery
* Patients on oral corticosteroid medication
* Patients on aspirin therapy < 7 days prior to operation

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2003-01; Study Completion 2005-06

PRIMARY OUTCOMES:
Comparison of the number of extravasated leukocytes in the skin blisters pre- and post-operatively, in both the placebo and aprotinin treatment groups

SECONDARY OUTCOMES:
The activation status of the blister leukocytes and the level of soluble inflammatory mediators within the blister

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Taylor, MD, FRCS, Principal Investigator — Hammersmith Hospital Campus, Imperial College
Locations (1):
- Hammersmith Hospital, London, United Kingdom

REFERENCES:
- [Background] Yagnik DR, Evans BJ, Florey O, Mason JC, Landis RC, Haskard DO. Macrophage release of transforming growth factor beta1 during resolution of monosodium urate monohydrate crystal-induced inflammation. Arthritis Rheum. 2004 Jul;50(7):2273-80. doi: 10.1002/art.20317. PMID 15248227
- [Background] Philippidis P, Mason JC, Evans BJ, Nadra I, Taylor KM, Haskard DO, Landis RC. Hemoglobin scavenger receptor CD163 mediates interleukin-10 release and heme oxygenase-1 synthesis: antiinflammatory monocyte-macrophage responses in vitro, in resolving skin blisters in vivo, and after cardiopulmonary bypass surgery. Circ Res. 2004 Jan 9;94(1):119-26. doi: 10.1161/01.RES.0000109414.78907.F9. Epub 2003 Dec 1. PMID 14656926